CLINICAL TRIAL: NCT02466022
Title: Does Single Dose Dexmedetomidine for Procedural Sedation Reduce Post-operative Pain in Total Knee Arthroplasty? A Randomized Control Study
Brief Title: Dexmedetomidine for Sedation in Total Knee Replacements
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Nirupan Vipulanathan, Anesthesiology Resident, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U of S BIO 15-76
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Post-operative Pain for Total Knee Arthroplasty
MeSH Terms: interventions — Dexmedetomidine; Bupivacaine; Saline Solution; normosol R; Fentanyl; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Patients will receive one 0.5ug/kg bolus of Dexmedetomidine over 10 minutes for sedation prior to spinal anesthetic (12.75mg of heavy Bupivicaine and 10ug of Fentanyl) and 0-4mg of Midazolam for rescue sedation
  Interventions: Drug: Dexmedetomidine; Drug: Bupivicaine; Drug: Normal Saline; Drug: Fentanyl; Drug: Midazolam
- Normal Saline (Placebo Comparator): Patients will receive 0.1cc/kg Normal Saline bolus delivered over 10 minutes for control arm prior to spinal anesthetic (12.75mg of heavy Bupivicaine and 10ug of Fentanyl) and 0-4mg of Midazolam for rescue sedation
  Interventions: Drug: Bupivicaine; Drug: Normal Saline; Drug: Fentanyl; Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Bolus dose prior to spinal anesthetic
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Bupivicaine — Intrathecal hyperbaric bupivicaine 12.75mg
  Other Names: Marcaine
Drug: Normal Saline — Bolus 0.1cc/kg Normal Saline over 10 min
  Other Names: Normosol
Drug: Fentanyl — Intrathecal Fentanyl 10ug
Drug: Midazolam — 0-4mg of IV Midazolam prn for rescue sedation
  Other Names: Versed

SUMMARY:
Dexmedetomidine has demonstrated benefits both in sedation, and post-operative pain control, with less respiratory depression than other common sedatives. Traditionally, dexmedetomidine has been used with a large loading dose and infusion, which has been known to cause dose-dependent negative side-effects (Abdallah et al., 2013). Single dose dexmedetomidine produces less negative side-effects, but still effective sedation and reduced post-operative pain (Jung et al., 2013). There is evidence for its benefits with general anesthesia but only a few studies exist investigating its benefits when administered for sedation purposes with spinal anesthesia, and no studies primarily examine post-operative opioid consumption. The investigators hypothesize that single dose dexmedetomidine for procedural sedation will reduce opioid consumption after total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
The investigators plan a randomized control trial.

Sample. Based on a literature and a previous study by the investigators team (RQHR #13-80/USask Bio #13-232), average reduction in opioid consumption for dexmedetomidine bolus and infusion is 50%. Less data exists for single dose. However two randomized control trials (Kaya et al., 2010; Hong et al., 2012) reduced consumption frequency by 55% and 45%, using 0.5ug/kg and 1.0ug/kg respectively. A meta-analysis demonstrated a mean difference of -10mg vs -21mg in opioid consumption for bolus studies vs bolus and infusion studies at 24 hours (Schnabel et. al 2013). A reduction of 50% was recently seen in a study conducted earlier by the investigators center at 24hours with a bolus and infusion (RQHR #13-80/USask Bio #13-232). An expected Patient Controlled Analgesia (PCA) consumption at 24hours for total knee arthroplasty is 27mg with a standard deviation of 19mg (Paul et. al, 2013). Using this information, it was decided 40% reduction in opioid consumption at 24hours could be expected and represent a clinically significant result. Subsequent power calculation required a sample size of 50 (25 per arm) to demonstrate a 40% reduction in opioid consumption at 24 hours, with a study power of 80% and P-value under 0.05.

Ethics. Ethics approval was obtained from the University of Saskatchewan Biomedical Research Ethics Board, and from the Regina Qu'Appelle Health Region Research Ethics Board.

Patients will be identified by one of the investigators through the daily surgical slate to which they already have access for patient care.

Informed written consent will be obtained from 50 patients on the Same-Day Admission Unit by one of the investigators not involved in the patient's care.

Randomization and Allocation. Following informed consent by one of the investigators, patients will be randomized into one of two groups based on a 1:1 ratio. Sealed envelopes will be prepared by the Department of Anesthesia's Research Coordinator using a web-based random number generator, and opened by a researcher (Dr. Maslany or Dr. Vipulananthan) independent of the clinical team. The drug will be prepared by a resident or nurse not involved in the patient's case; this staff member will vary depending on who is available when the need arises. Surgeons, anesthetists, ancillary staff and patients will be blinded to patient allocation.

Study Drug. The study drug (which does not require refrigeration) will be kept locked in the Anesthesia office at the Regina General Hospital. It has been arranged that Pharmacy will deliver the study drug in a batch, and the investigators will use a tracking sheet to account for the 25 vials that are required for the study. Both Dexmedetomidine and Normal saline are colorless and thus unrecognizable by either the patient or the anesthetist. There is no risk to the patient of delay in receiving midazolam at an appropriate time once the case is started. If the patient asks for more sedation at any time, it will be provided.

Procedure. Prior to entering the operating room, all patients will be familiarized with the Numerical Rating Scale (NRS) and instructed how to use patient controlled analgesia and instructions to press the PCA demand button if their NRS pain is 4 or greater. All patients will receive a 500cc bolus of lactated ringer's solution intravascular volume loading during spinal anesthetic delivery. Monitors include electrocardiography, non-invasive blood pressure measurement, pulse oximetry, and end-tidal carbon dioxide concentration with nasal prongs for monitoring respiration. Oxygen will be delivered at 3 litres per min.

Using a computer-generated randomization table by blinded staff, patients will be randomly allocated 1:1 to receive 0.5ug/kg of dexmedetomidine (experimental group) or same volume of normal saline (control group) over 10 min. The current standard of care, though variable, entails patients receiving a midazolam bolus for sedation during the operation, if the patient requests sedation. For patients who request sedation, a syringe of dexmedetomidine or saline will be run as a single dose infused over 10 minutes. However, a midazolam bolus (0-4 mg IV) will be available at the anesthetist's discretion to achieve a moderate sedation score as defined by the American Society of Anesthesiology.

Bupivicaine 0.75% 1.7cc (12.75mg) and fentanyl 10 micrograms will be administered intrathecally for analgesia 5 min after infusion has been completed.

The level of sensory block will be assessed, as per standard care, with pinpricks and ice cubes. Motor block will be assessed with a modified Bromage scale (0=no paralysis; 1=unable to raise extended leg; 2=unable to flex knee; 3=unable to flex ankle) (Bromage et al. 1964).

Rescue phenylephrine and ephedrine will be available to the anesthesiologist to use at their discretion for hypotension.

Patients will be discharged from post-anesthetic care unit, as per standard practice, once discharge criteria met as per modified Aldrete scoring system. For Total Knee Arthroplasty, the average PACU stay would be 45-60min. Patients will be kept until they meet the requirements of the modified Aldrete score and no longer, as per standard care.

Data collection. Baseline characteristics will be collected by Dr. Vipulananthan from the patients' charts, including: age, weight, height, sex, duration of surgery, baseline heart rate and blood pressure. Primary and secondary outcome measures will be collected, including: total morphine consumption at 6, 12, and 24hours, time to first morphine request, pain scores (Numerical Rating Scale) at 6, 12, and 24 hours at rest, intraoperative midazolam use, time of readiness of discharge from the post-anesthetic care unit, intraoperative and post-anesthetic care unit hemodynamics, duration of sensory and motor blockade by two-dermatome sensory regression, recovery of L2 dermatome sensation and knee flexion, adverse opioid effects of nausea, vomiting, pruritis, urinary retention, post-operative shivering, and patient satisfaction.

Analysis. Statistical methods will include multivariate analysis of variance and Mann-Whitney U-test to compare groups. There will be no crossover between groups and results will be analysed on an intention to treat basis. Sub-group analyses of Type II diabetic patients will be analyzed for insulin resistance. Statistical significance will be accepted at a probability level of under 0.05.

ELIGIBILITY:
Inclusion Criteria:

* adults over 18 years undergoing elective unilateral primary total knee arthroplasty under spinal anesthesia with an American Society of Anesthesiologists physical status class I to III.

Exclusion Criteria:

* will include contraindication to:

  * Dexmedetomidine,
  * morphine, or
  * Spinal Anesthesia,
* as well as anybody with chronic pain being treated by opioids prior to the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Total Morphine Consumption | 24 Hours
  mg of IV morphine administered via Patient Controlled Analgesia. Patient will be told to deliver morphine dose for pain =>4 from a numerical rating scale for pain from 0 to 10

SECONDARY OUTCOMES:
Morphine Consumption | 6, 12 and 24 hours, and time to first morphine request
  mg of IV morphine administered via Patient Controlled Analgesia. Patient will be told to deliver morphine dose for pain =>4 from a numerical rating scale for pain from 0 to 10
Pain | 6, 12 and 24 hours
  rated on a numerical rating scale for pain from 0 to 10
Intraoperative Midazolam | During the operation
  mg usage of IV midazolam for rescue sedation if patient requests more
Time of readiness of discharge from the post-anesthetic care unit | Immediately post-operation, average 1 hour
  minutes spent in PACU until criteria met by modified Aldrete Score
Intraoperative heartrate | During the operation
  Lowest heart rate recorded in beats per minute
Duration of sensory blockade two-dermatome sensory regression | During the operation, and immediately post-operation, average 1 hour
  Time in Minutes for recovery of 2 dermatomes of sensation
Adverse opioid effects of nausea | First 24 hours post-operation
  Binary yes/no if patient experienced nausea
Satisfaction | First 24 hours
  rated 0-4
Time to first morphine request | first 24 hours post-operation
  Time in minutes to first morphine request by patient
Intraoperative blood pressure | During the operation
  Lowest systolic blood pressure recorded in mmHg
Post-operative heartrate | Immediately after operation in PACU recovery, average 1 hour
  Lowest heartrate in PACU recorded in beats per minute
Post-operative blood pressure | Immediately after operation in PACU recovery, average 1 hour
  Lowest systolic blood pressure recorded in mmHg
Duration of Motor blockade | During the operation, and immediately post-operation, average 1 hour
  Time in minutes until patient regains knee flexion
Adverse opioid effect of vomiting | First 24 hours post-operation
  Binary yes/no if patient experienced vomiting
Adverse opioid effect of constipation | First 24 hours post-operation
  Binary yes/no if patient experienced constipation
Adverse anesthetic effect of shivering | Immediately after operation in PACU recovery, average 1 hour
  Binary yes/no if patient experienced shivering
Adverse opioid effect of pruritus | First 24 hours post-operation
  Binary yes/no if patient experienced pruritus
Adverse opioid effect of urinary retention | First 24 hours post-operation
  Binary yes/no if patient experienced urinary retention

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Maslany, MD, FRCPC, Principal Investigator — University of Regina
Locations (1):
- Regina Qu'Appelle Health Region, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Abdallah FW, Abrishami A, Brull R. The facilitatory effects of intravenous dexmedetomidine on the duration of spinal anesthesia: a systematic review and meta-analysis. Anesth Analg. 2013 Jul;117(1):271-8. doi: 10.1213/ANE.0b013e318290c566. Epub 2013 Apr 30. PMID 23632057
- [Background] Jung SH, Lee SK, Lim KJ, Park EY, Kang MH, Lee JM, Lee JJ, Hwang SM, Hong SJ. The effects of single-dose intravenous dexmedetomidine on hyperbaric bupivacaine spinal anesthesia. J Anesth. 2013 Jun;27(3):380-4. doi: 10.1007/s00540-012-1541-0. Epub 2013 Jan 10. PMID 23307164
- [Background] Kaya FN, Yavascaoglu B, Turker G, Yildirim A, Gurbet A, Mogol EB, Ozcan B. Intravenous dexmedetomidine, but not midazolam, prolongs bupivacaine spinal anesthesia. Can J Anaesth. 2010 Jan;57(1):39-45. doi: 10.1007/s12630-009-9231-6. Epub 2009 Dec 29. PMID 20039221
- [Background] Hong JY, Kim WO, Yoon Y, Choi Y, Kim SH, Kil HK. Effects of intravenous dexmedetomidine on low-dose bupivacaine spinal anaesthesia in elderly patients. Acta Anaesthesiol Scand. 2012 Mar;56(3):382-7. doi: 10.1111/j.1399-6576.2011.02614.x. Epub 2012 Jan 4. PMID 22220945
- [Background] Schnabel A, Meyer-Friessem CH, Reichl SU, Zahn PK, Pogatzki-Zahn EM. Is intraoperative dexmedetomidine a new option for postoperative pain treatment? A meta-analysis of randomized controlled trials. Pain. 2013 Jul;154(7):1140-9. doi: 10.1016/j.pain.2013.03.029. Epub 2013 Mar 27. PMID 23706726
- [Background] Paul JE, Nantha-Aree M, Buckley N, Cheng J, Thabane L, Tidy A, DeBeer J, Winemaker M, Wismer D, Punthakee D, Avram V. Gabapentin does not improve multimodal analgesia outcomes for total knee arthroplasty: a randomized controlled trial. Can J Anaesth. 2013 May;60(5):423-31. doi: 10.1007/s12630-013-9902-1. Epub 2013 Mar 12. PMID 23479393